CLINICAL TRIAL: NCT02140476
Title: Comparative Analysis Between A Bipolar Vessel Sealing and Cutting Device and the Tie and Suture Technique in Thyroidectomy: A Two Institution Randomized Clinical Trial
Brief Title: Comparative Analysis Between Bipolar Device and Conventional Tie & Suture Technique in Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: University of Sao Paulo (Other); Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: SCI-1151-13/13-1
Record Dates: First submitted 2014-05-09; First posted 2014-05-16 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Thyroid Goiter; Papillary Thyroid Cancer
Keywords: Thyroid goiter; Papillary thyroid cancer; Bipolar device; Sealing and cutting device; Thyroidectomy
MeSH Terms: conditions — Goiter; Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thyroid Goiter (Experimental): Benign thyroid disease with a nodule equal or lesser than 4 cm in diameter of any gender or ethnical origin. Half of these patients will undergo either bipolar or conventional thyroidectomy.
  Interventions: Device: Bipolar vessel sealing and cutting device; Procedure: Conventional thyroidectomy
- Papillary Thyroid Cancer (Active Comparator): Patients of any gender or ethnical origin with papillary thyroid cancer no greater than 4 cm in diameter. Half of these patients will undergo either bipolar or conventional thyroidectomy.
  Interventions: Device: Bipolar vessel sealing and cutting device; Procedure: Conventional thyroidectomy

INTERVENTIONS:
Device: Bipolar vessel sealing and cutting device — This device will be used in half of the patients with thyroid goiter and half of the patients with papillary thyroid cancer.
  Other Names: EnSeal® G2 Tissue Sealer
Procedure: Conventional thyroidectomy — Tie and suture technique. This device will be used in half of the patients with thyroid goiter and half of the patients with papillary thyroid cancer.

SUMMARY:
Bipolar sealing and cutting devices such as EnSeal® G2 Tissue Sealer are surgical instruments that use electrical powered diathermic energy to seal and transect tissue. These devices have shown high efficiency in a wide variety of open and laparoscopic general and gynecological surgical procedures.

The surgical performance of the EnSeal® has shown to be comparable to that of ultrasonic cutting devices in several studies. However, the efficacy of this instrument and in particular of new instruments such as the EnSeal® G2 Tissue Sealer has not been evaluated in thyroid surgery.

Our primary aim is to verify whether the EnSeal® performance is superior to the standard surgical technique for thyroidectomy in a randomized clinical trial on 2 different institutions.

DETAILED DESCRIPTION:
Background Bipolar sealing and cutting devices such as EnSeal® G2 Tissue Sealer are surgical instruments that use electrical powered diathermic energy to seal and transect tissue. These devices have shown high efficiency in a wide variety of open and laparoscopic general and gynecological surgical procedures.

The surgical performance of the EnSeal® has shown to be comparable to that of ultrasonic cutting devices in several studies. However, the efficacy of this instrument and in particular of new instruments such as the EnSeal® G2 Tissue Sealer has not been evaluated in thyroid surgery.

Primary Aim To verify whether the EnSeal® performance is superior to the standard surgical technique for thyroidectomy in a randomized clinical trial on 2 different institutions

Patients and Methods A total of 160 patients will be included in the study. They will be divided into two groups of 80 subjects. Patients will undergo thyroidectomy in each of the two institutions: The National Institute of Medical Sciences and Nutrition in Mexico City and the Clinical Hospital in Sao Paolo Brazil. Surgical indication for thyroidectomy will comprise benign or malign diseases.

Design A balanced randomized clinical trial design for assessing superiority in 2 institutions. Patients with benign or malign thyroid disease will be balanced a priori within the 2 groups of the study.

Sample Size Calculation The estimated number of cases was calculated based on potential differences in surgical time, which is the main outcome variable with the smallest difference to detect. Sample size was calculated assuming a hypothetical mean difference of 15 minutes with an 80% of statistical power, 95% of confidence, with a 5% of alpha error (Type I error) in a two-tied distribution hypothesis. Based on these assumptions a sample size of at least 75 subjects per group (arm) is necessary.

Institutional Review Board Evaluation The protocol will be submitted for evaluation to the Institutional Review Board of each institution and will have to be approved before enrolling the first patient. This protocol follows all institutional, governmental policies and medical regulations for clinical research in human beings.

Informed Consent and Ethical Considerations All patients will receive complete information about this protocol. After a brief explanation those who accept to be enrolled will need to sign an informed consent before surgery. It is necessary that two independent witness may sign too the informed consent. All included patients will be des-identified for keeping as anonymous all the records. A special registry number will be allocated for every included subject. All potential harms and risks will be minimized for maximize the benefits. This protocol will adhere to the respect of the human dignity, privacy and autonomy.

Trial Registry The trial will be registered in ClinicalTrials.gov before enrolling the first patient.

Randomization Each group of 80 patients will be divided into 2 subgroups, one with preoperative diagnosis of benign disease and other with preoperative diagnosis of papillary thyroid carcinoma. Four sets of 42 envelopes will be prepared for randomization. All four groups (one with a benign and the other with a malignant thyroid condition) will be independently randomized in both institutions at the time of induction of the anesthesia. In a total of 80 patients, the EnSeal® G2 Tissue Sealer will be used for thyroid resection once the sub-platysmal flaps have been developed and in the opposite group, the operation will be performed using the standard tie & suture technique by two experts.

Outcome Variables The primary outcomes will be operative time (minutes), blood loss (milliliters), loss of signal in laryngeal nerve monitoring, number of ligatures, pain intensity (score) and surgical complications (such as bleeding, hematoma, hypoparathyroidism, superior laryngeal nerve injury and recurrent laryngeal nerve palsy.

Operational Definitions

i. Operative Time Measured in minutes, starting at skin incision and ending with last closing suture of skin. Differences will be assessed using the t-student test.

ii. Blood Loss Measured in cc. Will be evaluated by weighting soaking sponges and collected blood through the aspiration cannula. Differences will be evaluated using the t-student test

iii. Loss of signal during continuous recurrent laryngeal nerve monitoring The number and time of loss or electromyography signaling of the recurrent laryngeal nerve will be recorded using continuous intraoperative neuro-monitoring and will be analyzed using the Fisher´s exact and the t-student tests

iv. Number of Ligatures: The number of ligatures placed on blood vessels will be recorded. Differences will be analyzed by the Fisher´s exact test or the Chi-squared test.

v. Pain Intensity All patients will receive a standard dose of pain medications. Pain will be assessed 12 and 24hs after surgery using a Visual Analogue Scale and pain medication dosing will be recorded. Differences will be analyzed using the t-test.

vi. Hypoparathyroidism Serum calcium, phosphorus, albumin and intact parathyroid hormone will be measured in every patient, 24 hours after surgery. Patients with a corrected calcium ≥7.5 mg/dl and no symptoms of hypocalcemia will receive no calcium supplements and no further blood tests will be obtained. In patients with symptoms (tingling trembling, parenthesis, tetanic, and cardiac manifestations) and/or corrected calcium <7.5 mg/dl. Ca supplements will be administered and calcium / phosphorus / albumin will be measured every 2 weeks until supplements have been weaned. In the case that hypocalcemia persisted for 3 months, calcium/ phosphorus / albumin will be measured monthly up to 6 months. Transient hypoparathyroidism will be considered if hypocalcemia recovers in less than 6 months and the diagnosis of permanent hypoparathyroidism will be established if hypocalcemia persists for more than 6 months. Differences will be analyzed using the Fisher´s exact test

vii. Recurrent Laryngeal Nerve Injury All patients will undergo preoperative and postoperative laryngoscopy the day after surgery. At the end of the operation, response of will be assessed by direct stimulation of the vagus nerve and the recurrent laryngeal nerve. Acoustic response and electrical amplitude will be recorded. In the absence of vocal cord abnormalities in the postoperative laryngoscopy, no further evaluations will be performed. If vocal cord paralysis or paresis were found in the postoperative laryngoscopy, patients will enter a voice rehabilitation program and subsequent laryngoscopies will be performed 2 weeks, 3 months and 6 months after surgery until recovery. Transient recurrent laryngeal nerve paralysis or paresis will be considered if vocal cord movement recovers in less than 6 months and the diagnosis of permanent vocal cord paralysis will be established if vocal cord abnormalities persist for more than 6 months. Differences will be analyzed using the Fisher´s exact test.

Data Collection and Analysis All the data obtained from the clinical files, laboratory exams and registers from the neuro-monitoring will be saved in an Excel sheet in a numerical range. All records and databases will be kept anonymous. Correspondence including private or personal data will be avoided. Statistical analysis will be performed with a commercially available software. Variable representation will be made by means of excel, SPSS or numbers.

All included variables will be analyzed based on their own scaling. Variable distribution will be tested before any statistical inference. Non-parametric analysis will be used in the case of a non-normal distribution. Any p value ≤5% or 0.05 (type I error) will be considered as statistically significant for a two-tied hypothesis.

Publication and Authorship Considerations Any data or result obtained from this study will be planed and discussed by the two principal investigators. Authorship inclusion will be based on the Vancouver Convention and the Friedman guidelines. An author must be qualified when he/she has participated on the conception and design of the study, acquisition of data, analysis and interpretation of the data.

Any partial or total publication or public presentation of the data of this protocol will require a previous authorization from the principal investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thyroid diseases amenable of surgical resection
2. Benign or malign thyroid disease
3. Thyroid nodules ≤ 4cm
4. Patients with any gender or ethnical origin
5. Adults patients with 18-65 years-old
6. Postoperative follow-up of at least 2 weeks
7. Patients competent to understand and sign the informed consent

Exclusion Criteria:

1. Patients with clinical or biochemical hyperthyroidism
2. Preoperative indication for lateral lymph node dissection (radical modified)
3. Presence of gross tracheal or laryngeal invasion with thyroid cancer
4. Preoperative vocal cord paralysis or laryngeal disease
5. Patients with bleeding disorders or using anticoagulants
6. Patients with advanced or undifferentiated thyroid cancer
7. Patients with secondary hyperparathyroidism or parathyroid disease
8. Patients who do not want to accept to participate in the study

Elimination Criteria:

1. Intraoperative indication of lateral lymph node dissection (radical modified)
2. Intraoperative requirement of any tracheal or laryngeal resection
3. Malfunction of the devices (EnSeal or neuro-monitoring)
4. Any intraoperative conditions of the patient that require to stop or modified the surgery
5. Incomplete records, laboratories or clinical follow-up
6. Patients from vulnerable populations or non-competent to understand or sign the informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Operative time and surgical safety | One year
  The primary outcomes will be operative time (minutes), blood loss (milliliters), transient and permanent hypoparathyroidism (calcium and PTH levels), loss of signal in laryngeal nerve monitoring, number of ligatures and pain intensity (EVA score).

SECONDARY OUTCOMES:
Surgical complications | one year
  The secondary outcome will determine if surgical complications (such as bleeding, hematoma, hypoparathyroidism, superior laryngeal nerve (SLN) injury and recurrent laryngeal nerve (RLN) palsy) are equivalent in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel F Herrrera, MD PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Erivelto Volpi, MD, Principal Investigator — Universidad de Sao Paulo
Locations (2):
- Hospital Das Clinicas, Universidad de Sao Paulo, São Paulo, São Paulo, Brazil
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Janssen PF, Brolmann HA, Huirne JA. Effectiveness of electrothermal bipolar vessel-sealing devices versus other electrothermal and ultrasonic devices for abdominal surgical hemostasis: a systematic review. Surg Endosc. 2012 Oct;26(10):2892-901. doi: 10.1007/s00464-012-2276-6. Epub 2012 Apr 27. PMID 22538684
- [Background] Person B, Vivas DA, Ruiz D, Talcott M, Coad JE, Wexner SD. Comparison of four energy-based vascular sealing and cutting instruments: A porcine model. Surg Endosc. 2008 Feb;22(2):534-8. doi: 10.1007/s00464-007-9619-8. Epub 2007 Dec 20. PMID 18097720
- [Background] Newcomb WL, Hope WW, Schmelzer TM, Heath JJ, Norton HJ, Lincourt AE, Heniford BT, Iannitti DA. Comparison of blood vessel sealing among new electrosurgical and ultrasonic devices. Surg Endosc. 2009 Jan;23(1):90-6. doi: 10.1007/s00464-008-9932-x. Epub 2008 May 16. PMID 18483824